CLINICAL TRIAL: NCT01155557
Title: Strength Capacity of Neck and Shoulder Muscles in Children and Adolescents 9-17 Years With Tension Type Headache and the Effect of Specific Strength-Training on Tension-Type Headache
Brief Title: The Effect of Specific Strength-Training on Tension-Type Headache in Children 9-17 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: The University Hospitals Centre for Nursing and Care Research, Copenhagen (Unknown); The Beckett-Fond (Unknown); The Fond of Jørgen Holm and Elisa F. Hansen (Unknown)
Responsible Party: Principal Investigator, Birte Tornoe, PhD, MSc, PT, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2009-081; 2009-41-3697 (Other: The Danish Data Council, Datatilsynet)
Record Dates: First submitted 2010-06-28; First posted 2010-07-02 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Tension-Type Headache
Keywords: Tension-Type Headache; Strength Capacity; Neck and Shoulder
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specific Strength Training (Active Comparator): 10 weeks of specific strength training of neck and shoulder muscles using elastic resistance.
  Interventions: Device: Specific Strength Training
- Lifestyle Counseling (Active Comparator): 10 weeks of counseling by nurse and physiotherapist in lifestyle changes.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Device: Specific Strength Training — 10 weeks of progressive specific strength training for neck and shoulder muscles.
  Other Names: A
  Arms: Specific Strength Training
Behavioral: Lifestyle Counseling — 10 weeks of counseling by nurse and physiotherapist in lifestyle changes.
  Other Names: B
  Arms: Lifestyle Counseling

SUMMARY:
This study aims at examining muscle strength capacity in neck and shoulder muscles in children and adolescents with and without tension-type headache, and furthermore examining the effect of a 10 week specific strength training programme for neck and shoulder muscles compared to a multi-disciplinary approach in 10 weeks.

DETAILED DESCRIPTION:
Frequent and chronic tension type headache are the most frequent pain illnesses in children with a prevalence of 0.5-7,6%. Frequent or daily headache leads to constraints in the child's life in relation to school and social activities.

The underlying pathophysiological mechanisms are not yet fully examined. In several studies in adults and in children it is found that the shoulder muscles are tense and tender, but it is not known whether this phenomenon is primary or secondary to tension-type headache. A decrease in muscle capacity is furthermore found in studies. We therefore aim at examining parameters for muscle function in order to compare the differences between children with and without headache, and at examining the effect of a 10 week progressive specific strength training programme on headache compared to an in time comparable multidisciplinary intervention based on lifestyle counseling.

ELIGIBILITY:
Inclusion Criteria:

* primary tension-type headache with no more than one episode of migraine pr. month

Exclusion Criteria:

* post-trauma headache
* co-morbidity

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Headache | At baseline
  Number of headache days/ 4 weeks. Mean VAS Score (pain)/4 weeks.
Muscle Capacity | At baseline
  Neck and shoulder muscle function variables:
  MVC(maximal voluntary static capacity). RFD(rate of force development). FS (Force-steadiness).
Headache | After the 10 weeks intervention programme
  Number of headache days/ 4 weeks. Mean VAS Score (pain)/4 weeks.
Headache | At 3 months follow up.
  Number of headache days/ 4 weeks. Mean VAS Score (pain)/4 weeks.
Muscle Capacity | After the 10 weeks intervention programme
  Neck and shoulder muscle function variables:
  MVC(maximal voluntary static capacity). RFD(rate of force development). FS(Force-steadiness).
Muscle Capacity | At 3 months follow up.
  Neck and shoulder muscle function variables:
  MVC(maximal voluntary static capacity). RFD(rate of force development). FS(Force-steadiness).

SECONDARY OUTCOMES:
TTS | At baseline
  Total Tenderness Score ( palpation of percranial tenderness).
Physical fitness | At baseline
  Submaximal ergometer bicycle test
TTS | After the 10 weeks intervention programme
  Total Tenderness Score ( palpation of pericranial tenderness).
TTS | At 3 months follow up.
  Total Tenderness Score ( palpation of pericranial tenderness).
Physical fitness | After the 10 weeks intervention programme
  Submaximal ergometer bicycle test
Physical fitness | At 3 months follow up.
  Submaximal ergometer bicycle test

CONTACTS AND LOCATIONS:
Overall Officials: Birte Tornøe, PhD,MSc,PT, Principal Investigator — Children's Headache Clinic, Herlev University Hospital, 2730 Herlev, Copenhagen-DK
Locations (1):
- Birte Tornøe, Copenhagen, Herlev, Denmark